CLINICAL TRIAL: NCT00728754
Title: A Prospective, Randomized-controlled Multicenter Study of the Osseotite Certain Lateralized Implant in Short-span Fixed Bridge Cases for Preservation of Crestal Bone
Brief Title: A Study of Certain Prevail Implants Used for the Preservation of Crestal Bone in Short Fixed Bridge Cases.
Acronym: Cliffhanger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2301x
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Results first posted 2011-11-17 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2022-03

CONDITIONS: Partial Edentulism; Tooth Disease
Keywords: dental implants; Osseotite Certain Prevail; Lateralized; non-lateralized; Osseotite Certain; multicenter; randomized; clinical study; partial edentulism; single stage; early loading; crestal bone level; short fixed bridge
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dental implant Osseotite Prevail (Experimental): Dental implant with lateralized design
  Interventions: Device: Dental implant Osseotite Prevail
- Dental implant Osseotite (Active Comparator): Dental implant without the lateralized design
  Interventions: Device: Dental implant Osseotite

INTERVENTIONS:
Device: Dental implant Osseotite Prevail — Root form titanium dental implant
  Other Names: Osseotite; Prevail
  Arms: Dental implant Osseotite Prevail
Device: Dental implant Osseotite — root form titanium dental implant
  Other Names: Osseotite
  Arms: Dental implant Osseotite

SUMMARY:
This prospective, randomized study will evaluate the performance of the Osseotite Certain Prevail implant when compared to that of the non-lateralized version of the implant.

Study (null) hypothesis: the crestal bone changes that take place after placement and loading of the Osseotite lateralized implants will be the same as for a similar but non-lateralized Osseotite Certain implant.

DETAILED DESCRIPTION:
This is a prospective, randomized, longitudinal study in which qualified patients with partial edentulism will receive a short-fixed bridge restoration. Each implant site is randomized to receive either the Osseotite Certain Lateralized (test) or the Osseotite Certain Non-lateralized (control). All implants will receive a temporary prosthesis after two months of placement. Enrollment will include up to 20 patients (approximately 60 implants per center) at each participating study center.

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex and any race greater than 18 years of age
* patients for whom a decision has already been made to use dental implants for treating an existing condition specifically: A partially edentulous short-span fixed case of less than 4 implants in the maxilla or mandible; the prosthesis may be anterior, posterior, or transitionally anterior-posterior; no cantilevers allowed but one interior crown may be a pontic
* patients must be physically able to tolerate conventional surgical and restorative procedures
* patients must agree to be evaluated for each study visit, especially the yearly follow-up visits

Exclusion Criteria:

* patients with active infection or severe inflammation in the areas intended for implant placement
* patients with a >10 cigarette per day smoking habit
* patients with uncontrolled diabetes mellitus
* patients with metabolic bone disease
* patients who have had treatment with therapeutic radiation to the head within the past 12 months
* patients in need of allogenic bone grafting a the site of the intended study implant
* patients who are pregnant at the screening visit
* patients with evidence of severe para-functional habits such as bruxing or clenching
* patients with cantilevers and more than one pontic per bridge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-03; Primary Completion 2007-07 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold Baumgarten, DMD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 120 patients were enrolled across all centers, with enrollment efforts beginning in February 2005. Enrollment period remained open until June 2006. Two participating sites were Universities and four were private practices.
Pre-assignment Details: Pre-treatment included a screening visit (enroll those meeting all inclusion criteria), signing informed consent, and pre-surgical data collection.Patients returned for implant placement surgery, followed by temporary prosthesis placement at 2 months.
Groups:
- Osseotite Certain Prevail Implant: Patients with dental implant with internal connection and expanded, lateralized design at coronal portion
- Osseotite Certain Implant: Patients with dental implant with internal connection and without the lateralized expanded platform design
Period: Implant Placement Surgery
Arm/Group | Osseotite Certain Prevail Implant | Osseotite Certain Implant
Started | 29 (Individual test implant units is 75) | 32 (Individual control implant units is 78)
Completed | 29 (Individual test implant units completed = 75) | 32 (Individual control implant units completed = 78)
Not Completed | 0 | 0
Period: Permanent Prosthesis Placement
Arm/Group | Osseotite Certain Prevail Implant | Osseotite Certain Implant
Started | 29 (Individual test implant units is 75) | 32 (Individual control implant units is 78)
Completed | 25 (Individual test implant units completed = 66) | 28 (Individual control implant units completed = 68)
Not Completed | 4 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 3 | 3
Period: One Year Post Placement Follow-up
Arm/Group | Osseotite Certain Prevail Implant | Osseotite Certain Implant
Started | 25 (individual test implant units is 66) | 28 (individual control implant units is 68)
Completed | 24 (individual test implant units completing is 65) | 28 (individual control implant units completed= 68)
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Two Year Post Placement Follow-up
Arm/Group | Osseotite Certain Prevail Implant | Osseotite Certain Implant
Started | 24 (individual test implant units is 65) | 28 (individual control implant units is 68)
Completed | 24 (individual test implant units completed= 65) | 28 (individual test implant units completed= 68)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Osseotite Certain Prevail Implant | Osseotite Certain Implant | Total
Number analyzed (Participants) | 29 | 32 | 61
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 21 | 39
  >=65 years | 11 | 11 | 22
Sex/Gender, Customized [Number; unit: participants]
  Female | 14 | 15 | 29
  Male | 15 | 17 | 32
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14
  Italy | 15 | 15 | 30
  Sweden | 5 | 4 | 9
  Australia | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Crestal Bone Regression (Amount of Bone Measured) Around Each Implant Unit
Description: Millimeters of crestal bone observed and measured in a radiograph of each study implant is measured and averaged to obtain the mean crestal bone loss or gain for each implant unit.
Time Frame: 1 year
Population: population analyzed was all patients receiving implants enrolled in the study, those reported here actually represent the number of implants being followed at the 12 month follow-up time point (time of analysis).
Measure: Mean (Standard Error); unit: millimeters
Units Other Than Participants: implants
Arm/Group | Osseotite Certain Prevail Implant | Osseotite Certain Implant
Number analyzed (Participants) | 24 | 28
Number analyzed (implants) | 65 | 68
millimeters | -0.7440 (0.1881) | -0.8445 (0.1439)

2. Secondary Outcome: Osseous Integration
Time Frame: four years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events are collected and reported from day 1 of the study to present, 4 years of study duration to date.
Description: Adverse event data is collected by patient questioning and visual examination of patient's mouth each study event visit.
Arm/Group | Osseotite Certain Prevail Implant | Osseotite Certain Implant
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/32
Other Adverse Events (participants affected / at risk) | 5/29 | 5/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osseotite Certain Prevail Implant (N=29) | Osseotite Certain Implant (N=32)
Loss of integration of implant (Surgical and medical procedures) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall furnish SPONSOR with a copy of any proposed publication thirty (30) days prior to submission for publication for review and comment. SPONSOR may request PI to delay publishing such proposed publication for a maximum of an additional sixty (60) days in order to protect the potential patentability of any invention described therein.